CLINICAL TRIAL: NCT01089218
Title: The Impact of Antibiotic Prophylaxis on Incidence of Post-bronchoscopy Fever and Change of Serum Cytokines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Deog Kyeom Kim, MD, Seoul Metropolitan Government, Seoul National University Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: postFB fever
Record Dates: First submitted 2010-03-14; First posted 2010-03-18 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Fever; Pneumonia
Keywords: bronchoscopy; post-bronchoscopy fever; pneumonia; cytokines; amoxicillin/clavulanate; prophylaxis
MeSH Terms: conditions — Fever; Pneumonia | interventions — Amoxicillin; Clavulanic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): control without intervention
  Interventions: Drug: control
- Amoxicillin/clavulanate (Active Comparator)
  Interventions: Drug: oral amoxicillin/clavulanate 1g (875/125mg)

INTERVENTIONS:
Drug: oral amoxicillin/clavulanate 1g (875/125mg) — oral amoxicillin/clavulanate 1g (875/125mg) on the day of the procedure 30 minutes prior to the FB
  Other Names: prophylaxis group
  Arms: Amoxicillin/clavulanate
Drug: control — no intervention with the same procedure of FB
  Arms: control

SUMMARY:
Fever can develop after fiberoptic bronchoscopy (FB) in about 2.5 - 16 % of adult patients. We evaluated the impact of oral amoxicillin/clavulanate (AC) on incidence of postbronchoscopic fever and pneumonia.

DETAILED DESCRIPTION:
For the population being undergone with bronchoscopy, the clinical signs and procedural measures for complication of bronchoscopy and cytokines will be checked.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or older) who underwent FB

Exclusion Criteria:

* concurrent treatment with antibiotics or systemic corticosteroid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The incidence of fever | 24 hr after bronchoscopy
  time frame for body temperature 24hr before and after bronchoscopy every 4hrs

SECONDARY OUTCOMES:
change of serum cytokines level | before bronchoscopy and 24hr after bronchoscopy
  Time frame for cytokine measurement 24hr before brochoscopy - 1hr after bronchosocpy - 24hr after brochoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Deog Kyeom Kim, MD., Study Director — Seoul Metropolitan Government, Seoul National University Boramae Medical Center, 39 Boramae-Gil, Dongjak-Gu, Seoul, Republic of Korea 156-707.

REFERENCES:
- [Derived] Park JS, Lee CH, Yim JJ, Yang SC, Yoo CG, Chung HS, Kim YW, Han SK, Shim YS, Kim DK. Impact of antibiotic prophylaxis on postbronchoscopy fever: a randomised controlled study. Int J Tuberc Lung Dis. 2011 Apr;15(4):528-35. doi: 10.5588/ijtld.10.0386. PMID 21396214